CLINICAL TRIAL: NCT07209631
Title: Is Lipoprotein-a Just a Lipid Marker or a Predictor for the Severity of Coronary Lesions in Aortic Valve Sclerosis Patients?
Brief Title: Serum Lipoprotein-a as a Marker of Severity of Coronary Artery Disease in Aortic Valve Sclerosis Patients
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Remon Saleh Adly, Lecturer of Cardiovascular, Faculty of Medicine, Sohag University, Sohag, Egypt., Sohag University
Other Study IDs: Soh-Med-24-09-5PD
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Serum; Lipoprotein(A); Severity; Coronary Artery Disease; Aortic Valve Sclerosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with chest pain and/or dyspnea were diagnosed provisionally as having coronary artery disease.
  Interventions: Other: Serum Lipoprotein-a level

INTERVENTIONS:
Other: Serum Lipoprotein-a level — A venous blood sample was taken from each patient a month or so after discharge to check their Lp (a) levels. The samples were centrifuged for 10 minutes at 2-8 °C, after which the serum was divided into aliquots and stored at -20 ° C.

SUMMARY:
This work aimed to evaluate the association of serum level of Lp(a) with the severity of coronary artery disease (CAD) in aortic valve sclerosis (AVS) patients.

DETAILED DESCRIPTION:
Aortic valve sclerosis (AVS) has a prevalence of 2% to 7% in the population above 65 years of age. In industrialized countries, aortic valve sclerosis is most frequently caused by progressive calcification and degeneration of the aortic cusps.

Coronary artery disease (CAD) is the most significant single cause of death in the world. In developed countries, more than 25% of all deaths in persons older than 35 years are due to CAD. More than half of acute myocardial infarctions occur without previous history or symptoms of CAD.

In recent years, there has been a special emphasis on lipoprotein(a) (Lp(a)), a significant, causal, and nonmodifiable predictor of valvular outcomes and CAD in the general population

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* Patients with chest pain and/or dyspnea were diagnosed provisionally as having coronary artery disease.

Exclusion Criteria:

* Aortic stenosis.
* Aortic prosthesis.
* Untreated hypothyroidism.
* Severe chronic kidney failure.
* Administration of anti-inflammatory or immunosuppressive drugs.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective cohort study was carried out on 100 patients. The study was done after approval from the local Ethics Committee (Under the Declaration of Helsinki). Informed written consent was obtained from the patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of significance of coronary lesions | 1 month post-procedure
  Incidence of significance of coronary lesions in relation to lipoprotein (a) level was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.